CLINICAL TRIAL: NCT05495009
Title: Birth Journey Through Virtual Reality :Pain, Anxiety and Birth Perception
Brief Title: Virtual Reality, Labor Pain, Anxiety, Birth Perception
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abant Izzet Baysal University (Other)
Responsible Party: Principal Investigator, Mervenur BÖYÜK, Research Assistant, Abant Izzet Baysal University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: İBDH-KDÜ-MB-01
Record Dates: First submitted 2022-07-06; First posted 2022-08-10 (Actual); Last update posted 2022-08-10 (Actual); Status verified 2022-08

CONDITIONS: Labor Pain; Anxiety
Keywords: labor; pain; anxiety; birth perception; virtual reality
MeSH Terms: conditions — Labor Pain; Anxiety Disorders; Pain

STUDY DESIGN:
Intervention Model Description: Randomized controlled experimental research
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of care (No Intervention): Introductory information form (IIF), labor follow-up form (FFL) and VAS-P, VAS-A were filled in the latent phase (1-3 cm). At the beginning of the active (4 cm) and transitional phases (8 cm), FFL, VAS-P and VAS-A were filled and no intervention was applied. 20 min in active phase. then, FFL, VAS-P and VAS-A were filled after 10 min in the transition phase. The Perception of Birth Scale is filled after birth.
- Standard of care+ virtual reality glasses (Experimental): Introductory information form (IIF), labor follow-up form (FFL) and VAS-P, VAS-A were filled in the latent phase (1-3 cm). At the beginning of the active (4 cm) and transitional phases (8 cm), after filling FFL, VAS-P and VAS-A, video was watched with virtual reality glasses. 20 minutes in active phase after watching the video. then, FFL, VAS-P and VAS-A were filled after 10 min in the transition phase. After the birth, the Perception of Birth Scale and Virtual Reality Satisfaction Form were filled.
  Interventions: Other: Standard of care+virtual reality glasses

INTERVENTIONS:
Other: Standard of care+virtual reality glasses — At the beginning of the active and transitional phases of labor, videos were watched with virtual reality glasses.
  Arms: Standard of care+ virtual reality glasses

SUMMARY:
The research was carried out in a randomized controlled trial to determine the effect of using virtual reality glasses on labor pain, anxiety, and labor perception of pregnant women. 60 pregnant women participated in the study at the Maternity and Children's Hospital located in the city center of Bolu. The data were collected via Introductory information form, Visual Comparison Scale-Pain, Visual Comparison Scale-Anxiety, labor follow-up form, Mother's Perception of Birth Scale, and virtual reality satisfaction evaluation form. Number, percentage, mean, standard deviation, Pearson chi-square, t-test for both groups were used to evaluate the data via the SPSS program. Statistical significance was accepted as p<0.05. Pregnant women in the experimental and control groups were found to be homogeneous in terms of sociodemographic and obstetric characteristics (p>0.05). At the beginning of labor, both pregnant groups showed similar score of the mean pain and anxiety(p>0.05). After applying 20 minutes in the active phase and 10 minutes in the transitional phase, the mean pain and anxiety scores of the experimental group were found to be lower, and this difference was found to be statistically significant(p<0.001). In the postpartum period, it was determined that the birth Perception Scale mean scores of the groups were similar. 90% of the pregnant women reported that they were satisfied with the virtual reality application and 93% of them reported that they would recommend this application. As a result, the use of virtual reality during birth reduces pain and anxiety at birth but does not affect the perception of birth.

DETAILED DESCRIPTION:
Childbirth is one of the important experiences in a woman's life and this experience is affected by subjective, psychological and physiological processes. While birth is a positive life experience for some women , it is a traumatic and negative experience for others .

One of the factors that most affect women who experience many emotions together during the birth process is labor pain. The perception and severity of labor pain, which is part of the normal process, varies from person to person. In the literature, it has been shown that 50-52% of women experience severe labor pain. Severe labor pain may be associated with decreased uteroplacental perfusion, prolongation of labor and labor with intervention, postpartum depression and anxiety by causing an increase in maternal catecholamine levels. This leads to a prolonged hospital stay, difficulty in performing basic activities, and consequently a negative birth experience It also leads women who want to avoid pain to prefer cesarean delivery instead of vaginal delivery.

The birth process is also an important source of anxiety in women. Studies have shown that women experience moderate anxiety about childbirth. It is known that anxiety experienced at birth affects the health of the mother, fetus and newborn negatively and increases the severity of labor pain. Pain that comes at frequent and intense intervals increases the anxiety level of the woman, leading to increased tension in the pelvic muscles, fatigue, and inadequate coping with pain . There is a two-way relationship between anxiety and pain in childbirth, and this vicious cycle between anxiety and pain negatively affects the course of labor, reduces the self-confidence of the pregnant woman and causes her to feel helpless and unsuccessful.

Pain and anxiety are important factors affecting birth perception and birth outcomes. Effective management of pain and anxiety at birth for a positive birth experience is among the main goals of obstetric care. The most effective strategies for a positive birth experience; It has been reported that creating a positive birth environment, supporting women during childbirth, intrapartum care with minimal intervention, preparation for childbirth, relaxation and pain relief applications .

Pharmacological and non-pharmacological methods are used to effectively cope with pain at birth. Pharmacological methods require attention in their use because of their side effects, application limitations, and uncertainties of their effects on the mother and fetus .

The use of non-pharmacological methods, which are easy to apply, safe, and have various advantages in ensuring active participation and cooperation of women in the birth process, without using any medication, is becoming more common in pain management. Studies have emphasized that non-pharmacological methods reduce pain and anxiety levels during the birth process, increase maternal satisfaction at birth, and strengthen mother-infant communication.

Distraction, focusing and relaxation by daydreaming are among the commonly used non-pharmacological methods in reducing pain. However, since dreaming and daydreaming can be difficult during the birth process, it is recommended to use applications that will facilitate this . For this purpose, virtual reality glasses have been used in recent years. With these glasses, a visual experience environment is created through three-dimensional videos by creating a real-like virtual world for individuals.

It has been shown that the clinical use of virtual reality glasses, which can be used in many areas, is useful and reliable. These glasses are used in children during painful invasive procedures, acute and chronic pain management, burn treatments, preoperative anxiety, psychiatric diagnosis and treatment interventions, physical therapy and rehabilitation applications are used.

Although virtual reality has been shown to be an effective method in the management of pain and anxiety, studies showing its effect on pain at birth and anxiety are limited. Based on these data, in this study, it was aimed to determine the effect of the video watched by using virtual reality glasses during labor on labor pain, anxiety and labor perception of pregnant women.

Research Hypotheses H0 : Watching video with virtual reality glasses has no effect on labor pain, anxiety and birth perception.

H1: Watching video with virtual reality glasses has an effect on labor pain. H2: Watching video with virtual reality glasses has an effect on anxiety at birth.

H3: Watching a video with virtual reality glasses has an effect on birth perception.

ELIGIBILITY:
Inclusion Criteria:

* Able to communicate verbally
* Between the ages of 18-35
* No pregnancy-related risk diagnosis,
* Primiparous,
* Vaginal delivery planned,
* Gestational week is between 37-42,
* Single, live fetus and head presentation,
* In the latent phase (1-3 cm) on admission to the delivery room,
* Not having any dystocia that may affect the duration of labor (placental dystocia, pelvic dystocia, etc.).
* No induction,
* No epidural anaesthesia.
* Pregnant women without vision and hearing problems were included in the study.

Exclusion Criteria:

* Refusing to participate in the research,
* Diagnosed with risky pregnancy,
* Watching the video in active phase for less than 20 minutes
* Watching the video in transition phase for less than 10 minutes
* Cesarean section
* Pregnant women who used any pharmacological analgesia were not included in the study.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — The study was carried out with women in accordance with the subject of the study.
Enrollment: 60 (Actual)
Dates: Start 2021-06-21 (Actual); Primary Completion 2021-12-12 (Actual); Study Completion 2021-12-12 (Actual)

PRIMARY OUTCOMES:
pre-intervention pain at the start of the active phase was assessed by Visual Analogue Scale-Pain (VAS-P) | It was applied before the intervention was performed when the cervical opening was 4 cm.
  The scale is a 10 cm ruler that represents painlessness at one end (0=no pain) and the most severe pain (10=severe pain) at the other end. The patient is asked to put a line or mark on the point representing the intensity of pain. The part from the "no pain" point to the point marked by the participant is measured in mm and the value found indicates the patient's pain level.
post-intervention pain at the start of the active phase was assessed Visual Analogue Scale-Pain (VAS-P) | It was applied after the intervention was performed when the cervical opening was 4 cm.
  The scale is a 10 cm ruler that represents painlessness at one end (0=no pain) and the most severe pain (10=severe pain) at the other end. The patient is asked to put a line or mark on the point representing the intensity of pain. The part from the "no pain" point to the point marked by the participant is measured in mm and the value found indicates the patient's pain level.
pre-intervention anxiety at the start of the active phase was assessed by Visual Analogue Scale-Anxiety (VAS-A) | It was applied before the intervention was performed when the cervical opening was 4 cm.
  The scale is a 10 cm ruler representing the absence of anxiety (0 = no anxiety) at one end and the most severe anxiety (10 = severe anxiety) at the other end. The patient is asked to put a line or mark on the area showing the level of anxiety. The part from the no anxiety point to the point marked by the patient is measured in mm and the value found indicates the patient's anxiety level.
post-intervention anxiety at the start of the active phase was assessed by Visual Analogue Scale-Anxiety (VAS-A) | It was applied after the intervention was performed when the cervical opening was 4 cm.
  The scale is a 10 cm ruler representing the absence of anxiety (0 = no anxiety) at one end and the most severe anxiety (10 = severe anxiety) at the other end. The patient is asked to put a line or mark on the area showing the level of anxiety. The part from the no anxiety point to the point marked by the patient is measured in mm and the value found indicates the patient's anxiety level.
pre-intervention pain at the start of the transition phase was assessed by Visual Analogue Scale-Pain (VAS-P) | It was applied before the intervention was performed when the cervical opening was 8 cm.
  The scale is a 10 cm ruler that represents painlessness at one end (0=no pain) and the most severe pain (10=severe pain) at the other end. The patient is asked to put a line or mark on the point representing the intensity of pain. The part from the "no pain" point to the point marked by the participant is measured in mm and the value found indicates the patient's pain level.
post-intervention pain at the start of the transition phase was assessed by Visual Analogue Scale-Pain (VAS-P) | It was applied after the intervention was performed when the cervical opening was 8 cm.
  The scale is a 10 cm ruler that represents painlessness at one end (0=no pain) and the most severe pain (10=severe pain) at the other end. The patient is asked to put a line or mark on the point representing the intensity of pain. The part from the "no pain" point to the point marked by the participant is measured in mm and the value found indicates the patient's pain level.
pre-intervention anxiety at the start of the transition phase was assessed by Visual Analogue Scale-Anxiety (VAS-A) | It was applied before the intervention was performed when the cervical opening was 8 cm.
  The scale is a 10 cm ruler representing the absence of anxiety (0 = no anxiety) at one end and the most severe anxiety (10 = severe anxiety) at the other end. The patient is asked to put a line or mark on the area showing the level of anxiety. The part from the no anxiety point to the point marked by the patient is measured in mm and the value found indicates the patient's anxiety level.
post-intervention anxiety at the start of the transition phase was assessed by Visual Analogue Scale-Anxiety (VAS-A) | It was applied after the intervention was performed when the cervical opening was 8 cm.
  The scale is a 10 cm ruler representing the absence of anxiety (0 = no anxiety) at one end and the most severe anxiety (10 = severe anxiety) at the other end. The patient is asked to put a line or mark on the area showing the level of anxiety. The part from the no anxiety point to the point marked by the patient is measured in mm and the value found indicates the patient's anxiety level.
birth perception in the postpartum period was assessed by Mother's Perception of Birth Scale | postpartum 4 hour
  The Mother's Perception of Birth Scale, which evaluates the experiences and perceptions of mothers at the time of birth, was developed by Fawcett and Knauth (144). The Turkish validity and reliability study of the scale was carried out by Güngör and Beji (2007). Experiences at the time of birth (7 items; 3, 5, 6, 8, 15, 17, 18), experiences during the pain period of labor (7 items; 1, 2, 4, 7, 9, 10, 16), postpartum (4 items) It consists of a total of 5 sub-dimensions and 25 items, namely; 22, 23, 24, 25), partner involvement (4 items; 11,12,20,21) and awareness (3 items; 13,14,19). Each item is scored from 1 to 5 in the Mother's Perception of Birth Scale. It is evaluated as 1-Not at all, 2-A little, 3-Moderate, 4-Very, 5-Very much. Since the questions 15-16-17-18-19 of the scale contain negative statements, scoring is done in reverse for these questions.

SECONDARY OUTCOMES:
pre-intervention systolic blood pressure (mmHg) at the start of the active phase was assessed. | It was applied before the intervention was performed when the cervical opening was 4 cm.
  systolic blood pressure, measures the pressure in your arteries when your heart beats. Measurements were made with a blood pressure monitor.
post-intervention systolic blood pressure (mmHg) at the start of the active phase was assessed. | It was applied after the intervention was performed when the cervical opening was 4 cm.
  systolic blood pressure, measures the pressure in your arteries when your heart beats. Measurements were made with a blood pressure monitor.
pre-intervention diastolic blood pressure (mmHg) at the start of the active phase was assessed. | It was applied before the intervention was performed when the cervical opening was 4 cm.
  diastolic blood pressure, measures the pressure in your arteries when your heart rests between beats. Measurements were made with a blood pressure monitor.
post-intervention diastolic blood pressure (mmHg) at the start of the active phase was assessed. | It was applied after the intervention was performed when the cervical opening was 4 cm.
  diastolic blood pressure, measures the pressure in your arteries when your heart rests between beats. Measurements were made with a blood pressure monitor.
pre-intervention pulse (minute) at the start of the active phase was assessed. | It was applied before the intervention was performed when the cervical opening was 4 cm.
  The rhythmic dilation of an artery that results from beating of the heart. Measurements were made with a heart rate monitor.
post-intervention pulse (minute) at the start of the active phase was assessed. | It was applied after the intervention was performed when the cervical opening was 4 cm.
  The rhythmic dilation of an artery that results from beating of the heart. Measurements were made with a heart rate monitor.
pre-intervention respiration (minute) at the start of the active phase was assessed. | It was applied before the intervention was performed when the cervical opening was 4 cm.
  the inhaling of oxygen and the exhaling of carbon dioxide. is found by counting the number of breaths (how many times the chest rises).
post-intervention respiration (minute) at the start of the active phase was assessed. | It was applied after the intervention was performed when the cervical opening was 4 cm.
  the inhaling of oxygen and the exhaling of carbon dioxide. is found by counting the number of breaths (how many times the chest rises).
pre-intervention fetal heart rate (minute) at the start of the active phase was assessed. | It was applied before the intervention was performed when the cervical opening was 4 cm.
  Fetal heart rate was measured using a fetal Doppler device.
post-intervention fetal heart rate (minute) at the start of the active phase was assessed. | It was applied after the intervention was performed when the cervical opening was 4 cm.
  Fetal heart rate was measured using a fetal Doppler device.
pre-intervention contraction frequency (minute) at the start of the active phase was assessed. | It was applied before the intervention was performed when the cervical opening was 4 cm.
  Measurements were made using the NST device.
post-intervention contraction frequency (minute) at the start of the active phase was assessed. | It was applied after the intervention was performed when the cervical opening was 4 cm.
  Measurements were made using the NST device.
pre-intervention contraction duration (minute) at the start of the active phase was assessed. | It was applied before the intervention was performed when the cervical opening was 4 cm.
  Measurements were made using the NST device.
post-intervention contraction duration (minute) at the start of the active phase was assessed. | It was applied after the intervention was performed when the cervical opening was 4 cm.
  Measurements were made using the NST device.
pre-intervention contraction severity (minute) at the start of the active phase was assessed. | It was applied before the intervention was performed when the cervical opening was 4 cm.
  Measurements were made using the NST device.
post-intervention contraction severity (minute) at the start of the active phase was assessed. | It was applied after the intervention was performed when the cervical opening was 4 cm.
  Measurements were made using the NST device.
pre-intervention systolic blood pressure (mmHg) at the start of the transition phase was assessed. | It was applied before the intervention was performed when the cervical opening was 8 cm.
  systolic blood pressure, measures the pressure in your arteries when your heart beats. Measurements were made with a blood pressure monitor.
post-intervention systolic blood pressure (mmHg) at the start of the transition phase was assessed. | It was applied after the intervention was performed when the cervical opening was 8 cm.
  systolic blood pressure, measures the pressure in your arteries when your heart beats. Measurements were made with a blood pressure monitor.
pre-intervention diastolic blood pressure (mmHg) at the start of the transition phase was assessed. | It was applied before the intervention was performed when the cervical opening was 8 cm.
  diastolic blood pressure, measures the pressure in your arteries when your heart rests
post-intervention diastolic blood pressure (mmHg) at the start of the transition phase was assessed. | It was applied after the intervention was performed when the cervical opening was 8 cm.
  diastolic blood pressure, measures the pressure in your arteries when your heart rests
pre-intervention pulse (minute) at the start of the transition phase was assessed. | It was applied before the intervention was performed when the cervical opening was 8 cm.
  The rhythmic dilation of an artery that results from beating of the heart. Measurements were made with a heart rate monitor.
post-intervention pulse (minute) at the start of the transition phase was assessed. | It was applied after the intervention was performed when the cervical opening was 8 cm.
  The rhythmic dilation of an artery that results from beating of the heart. Measurements were made with a heart rate monitor.
pre-intervention respiration (minute) at the start of the transition phase was assessed. | It was applied before the intervention was performed when the cervical opening was 8 cm.
  the inhaling of oxygen and the exhaling of carbon dioxide. is found by counting the number of breaths (how many times the chest rises).
post-intervention respiration (minute) at the start of the transition phase was assessed. | It was applied after the intervention was performed when the cervical opening was 8 cm.
  the inhaling of oxygen and the exhaling of carbon dioxide. is found by counting the number of breaths (how many times the chest rises).
pre-intervention fetal heart rate (minute) at the start of the transition phase was assessed. | It was applied before the intervention was performed when the cervical opening was 8 cm.
  Fetal heart rate was measured using a fetal Doppler device.
post-intervention fetal heart rate (minute) at the start of the transition phase was assessed. | It was applied after the intervention was performed when the cervical opening was 8 cm.
  Fetal heart rate was measured using a fetal Doppler device.
pre-intervention contraction frequency (minute) at the start of the transition phase was assessed. | It was applied before the intervention was performed when the cervical opening was 8 cm.
  Measurements were made using the NST device.
post-intervention contraction frequency (minute) at the start of the transition phase was assessed. | It was applied after the intervention was performed when the cervical opening was 8 cm.
  Measurements were made using the NST device.
pre-intervention contraction duration (minute) at the start of the transiton phase was assessed. | It was applied before the intervention was performed when the cervical opening was 8 cm.
  Measurements were made using the NST device.
post-intervention contraction duration (minute) at the start of the transiton phase was assessed. | It was applied after the intervention was performed when the cervical opening was 8 cm.
  Measurements were made using the NST device.
pre-intervention contraction severity (minute) at the start of the transition phase was assessed. | It was applied before the intervention was performed when the cervical opening was 8 cm.
  Measurements were made using the NST device.
post-intervention contraction severity (minute) at the start of the transition phase was assessed. | It was applied after the intervention was performed when the cervical opening was 8 cm.
  Measurements were made using the NST device.

CONTACTS AND LOCATIONS:
Overall Officials: Mervenur BÖYÜK, Principal Investigator — Baibu
Locations (1):
- İzzet Baysal State Hospital, Obstetrics and Pediatrics Unit, delivery room service, Bolu, Center, Turkey (Türkiye)

REFERENCES:
- [Derived] Boyuk M, Citak Bilgin N. Childbirth Journey Through Virtual Reality: Pain, Anxiety and Birth Perception: A Randomized Controlled Trial. Res Nurs Health. 2025 Apr;48(2):179-189. doi: 10.1002/nur.22438. Epub 2025 Jan 3. PMID 39749486